CLINICAL TRIAL: NCT06592066
Title: Accuracy of Digital Intraoral Scanning With and Without Prefabricated Landmarks Versus Conventional Impression Technique for Mandibular Implant Supported Full-Arch Prosthesis
Brief Title: Digital Intraoral Scanning With and Without Prefabricated Landmarks Versus Conventional Impression Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Kirollos Sobhy Kamel Shanoudy, Associate Lecturer, Ain Shams University
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: FDASU-Rec ID022403
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dental Impression Technique

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Splinted Conventional Impression Technique (Active Comparator): Splinted open tray conventional impression technique will be used for the mandibular full-arch implants, utilizing medium body impression material.
  Interventions: Device: Splinted Open Top Tay Conventional Impression Technique
- Digital impression technique with scan bodies (Experimental): Digital impression technique will be employed for mandibular full-arch implants, using intraoral scanning with scan bodies to capture the implant positions.
  Interventions: Device: Digital Impression by using Intraoral Scanning of Scan Bodies
- Digital impression technique with scan bodies with Prefabricated Landmarks (Experimental): Digital impression technique will be employed for mandibular full-arch implants, using intraoral scanning with scan bodies with prefabricated landmarks to capture the implant positions.
  Interventions: Device: Digital Impression by using Intraoral Scanning of Scan Bodies with Prefabricated Landmarks

INTERVENTIONS:
Device: Digital Impression by using Intraoral Scanning of Scan Bodies — intraoral scanning will be used to capture the positions of full-arch mandibular implants with the aid of scan bodies.
  Arms: Digital impression technique with scan bodies
Device: Digital Impression by using Intraoral Scanning of Scan Bodies with Prefabricated Landmarks — intraoral scanning will be used to capture the positions of full-arch mandibular implants with the aid of scan bodies with prefabricated landmarks in place.
  Arms: Digital impression technique with scan bodies with Prefabricated Landmarks
Device: Splinted Open Top Tay Conventional Impression Technique — Splinted open-top tray conventional impression technique will be preformed by using medium body silicone impression material.
  Arms: Splinted Conventional Impression Technique

SUMMARY:
The aim of this clinical trial is to evaluate the accuracy of digital implant impressions with or without prefabricated landmarks between scan bodies compared to conventional impression technique in mandibular full-arch implant cases.

DETAILED DESCRIPTION:
Implant-supported full arch dental prostheses are crucial and reliable alternatives for individuals with missing teeth in their jaws. The initial phase in the production of implant-supported prostheses involves the impression-taking process. Inaccurate impressions can result in a misfit between the prosthesis and implant abutment, potentially causing both mechanical and biological complications that can adversely affect the long-term viability of the implants. Therefore, the precision of impressions is of utmost importance, particularly for prostheses supported by multiple implants.

The conventional approach to obtaining impressions for multiple implants involves the use of an open-tray technique, widely adopted in dental practice. In this method, impression copings are connected to prevent rotational movements, making it a preferable choice compared to the non-splinting technique. Nevertheless, this procedure is complex, less efficient, and demands considerable clinical expertise. It is advised for use by experienced dentists, as those lacking experience have shown a notably higher rate of unsuccessful outcomes when employing the splinting technique.6 Additionally, various factors, such as patients' pharyngeal reflex and the potential deformation of impression materials, can influence the accuracy of implant impressions in the conventional workflow.

With the advancement of computer-aided design/computer-aided manufacturing (CAD/CAM) and digital technologies, the intraoral scanner (IOS) has gained popularity for capturing implant positions. In clinical practice, IOSs are valued for their comfort, efficiency, and practicality. However, it's important to note that IOSs cannot completely replace traditional methods. When it comes to implant-supported fixed dental prostheses, intraoral scanners can effectively be used for single- and three-unit implant scanning.

In a study from 2020, Revell et al. recommended specific scanners, such as Primescan, for complete-arch implant impressions due to their low deviation values at the implant platform level. Nevertheless, the accuracy of older models of intraoral scanners may not be reliable when scanning edentulous spaces with long inter-implant distances or fully edentulous jaws, particularly in the hands of inexperienced operators.

Previous research has introduced custom-designed scan bodies featuring an extensional structure to achieve dependable digital full-arch implant impressions. Typically, these platforms necessitate the use of custom-made scan bodies or a secondary scan to obtain mucosal information. In this context, this study is conducted to present newly designed prefabricated landmarks between the scan bodies to offer a solution for digital scanning of a mandibular full-arch implant. Therefore, the aim of this study is to evaluate and compare the accuracy of digital intraoral scanning with or without prefabricated landmarks to conventional impression techniques in mandibular full-arch implant cases.

The null hypothesis posits that there would be no significant difference in accuracy between digital intraoral scanning with or without prefabricated landmarks between scan bodies and conventional impression techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients with completely edentulous mandible, non-smokers, 50-70 years in age, have Good oral hygiene and motivation.

Exclusion Criteria:

* patients with major systemic diseases that may affect osseointegration as uncontrolled diabetes mellitus, the need for extensive bone grafting in planned implant site, pregnancy, patients under bisphosphonate treatment, and limited mouth-opening for executing the guided implant surgery.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The accuracy of digital intraoral scanning of full-arch mandibular implants. | Baseline
  Improving digital intraoral scanning of mandibular full-arch implant cases will facilitate the impression procedure, omit the drawback of conventional impression, improve the passive fit, and address the biomechanical considerations of the final-full arch prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Ingy A. Talaat, PHD, Study Director — Ain Shams Univeristy; Noha H. Nawar, PHD, Study Director — Ain Shams Univeristy; Omar A. El-Sadat, PHD, Study Director — Ain Shams Univeristy; Omnia M. Refai, PHD, Study Director — Ain Shams Univeristy

REFERENCES:
- [Background] Papaspyridakos P, Mokti M, Chen CJ, Benic GI, Gallucci GO, Chronopoulos V. Implant and prosthodontic survival rates with implant fixed complete dental prostheses in the edentulous mandible after at least 5 years: a systematic review. Clin Implant Dent Relat Res. 2014 Oct;16(5):705-17. doi: 10.1111/cid.12036. Epub 2013 Jan 11. PMID 23311617
- [Background] Goodacre CJ, Bernal G, Rungcharassaeng K, Kan JY. Clinical complications with implants and implant prostheses. J Prosthet Dent. 2003 Aug;90(2):121-32. doi: 10.1016/S0022-3913(03)00212-9. PMID 12886205
- [Background] Pjetursson BE, Thoma D, Jung R, Zwahlen M, Zembic A. A systematic review of the survival and complication rates of implant-supported fixed dental prostheses (FDPs) after a mean observation period of at least 5 years. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:22-38. doi: 10.1111/j.1600-0501.2012.02546.x. PMID 23062125
- [Background] Papaspyridakos P, Chen CJ, Gallucci GO, Doukoudakis A, Weber HP, Chronopoulos V. Accuracy of implant impressions for partially and completely edentulous patients: a systematic review. Int J Oral Maxillofac Implants. 2014 Jul-Aug;29(4):836-45. doi: 10.11607/jomi.3625. PMID 25032763
- [Background] Papaspyridakos P, Gallucci GO, Chen CJ, Hanssen S, Naert I, Vandenberghe B. Digital versus conventional implant impressions for edentulous patients: accuracy outcomes. Clin Oral Implants Res. 2016 Apr;27(4):465-72. doi: 10.1111/clr.12567. Epub 2015 Feb 13. PMID 25682892
- [Background] Perez-Davidi M, Levit M, Walter O, Eilat Y, Rosenfeld P. Clinical accuracy outcomes of splinted and nonsplinted implant impression methods in dental residency settings. Quintessence Int. 2016;47(10):843-852. doi: 10.3290/j.qi.a36323. PMID 27284582
- [Background] Miyoshi K, Tanaka S, Yokoyama S, Sanda M, Baba K. Effects of different types of intraoral scanners and scanning ranges on the precision of digital implant impressions in edentulous maxilla: An in vitro study. Clin Oral Implants Res. 2020 Jan;31(1):74-83. doi: 10.1111/clr.13548. Epub 2019 Oct 28. PMID 31608509
- [Background] Nagata K, Fuchigami K, Okuhama Y, Wakamori K, Tsuruoka H, Nakashizu T, Hoshi N, Atsumi M, Kimoto K, Kawana H. Comparison of digital and silicone impressions for single-tooth implants and two- and three-unit implants for a free-end edentulous saddle. BMC Oral Health. 2021 Sep 23;21(1):464. doi: 10.1186/s12903-021-01836-1. PMID 34556111
- [Background] Revell G, Simon B, Mennito A, Evans ZP, Renne W, Ludlow M, Vag J. Evaluation of complete-arch implant scanning with 5 different intraoral scanners in terms of trueness and operator experience. J Prosthet Dent. 2022 Oct;128(4):632-638. doi: 10.1016/j.prosdent.2021.01.013. Epub 2021 Apr 6. PMID 33832761
- [Background] Tan MY, Yee SHX, Wong KM, Tan YH, Tan KBC. Comparison of Three-Dimensional Accuracy of Digital and Conventional Implant Impressions: Effect of Interimplant Distance in an Edentulous Arch. Int J Oral Maxillofac Implants. 2019 March/April;34(2):366-380. doi: 10.11607/jomi.6855. Epub 2018 Dec 5. PMID 30521661
- [Background] Lyu M, Di P, Lin Y, Jiang X. Accuracy of impressions for multiple implants: A comparative study of digital and conventional techniques. J Prosthet Dent. 2022 Nov;128(5):1017-1023. doi: 10.1016/j.prosdent.2021.01.016. Epub 2021 Feb 25. PMID 33640093
- [Background] Thanasrisuebwong P, Kulchotirat T, Anunmana C. Effects of inter-implant distance on the accuracy of intraoral scanner: An in vitro study. J Adv Prosthodont. 2021 Apr;13(2):107-116. doi: 10.4047/jap.2021.13.2.107. Epub 2021 Apr 27. PMID 34025959
- [Background] Resende CCD, Barbosa TAQ, Moura GF, Tavares LDN, Rizzante FAP, George FM, Neves FDD, Mendonca G. Influence of operator experience, scanner type, and scan size on 3D scans. J Prosthet Dent. 2021 Feb;125(2):294-299. doi: 10.1016/j.prosdent.2019.12.011. Epub 2020 Feb 27. PMID 32115221
- [Background] Huang R, Liu Y, Huang B, Zhang C, Chen Z, Li Z. Improved scanning accuracy with newly designed scan bodies: An in vitro study comparing digital versus conventional impression techniques for complete-arch implant rehabilitation. Clin Oral Implants Res. 2020 Jul;31(7):625-633. doi: 10.1111/clr.13598. Epub 2020 Apr 3. PMID 32181919
- [Background] Huang R, Liu Y, Huang B, Zhou F, Chen Z, Li Z. Improved accuracy of digital implant impressions with newly designed scan bodies: an in vivo evaluation in beagle dogs. BMC Oral Health. 2021 Dec 7;21(1):623. doi: 10.1186/s12903-021-01986-2. PMID 34876122
- [Background] Iturrate M, Eguiraun H, Solaberrieta E. Accuracy of digital impressions for implant-supported complete-arch prosthesis, using an auxiliary geometry part-An in vitro study. Clin Oral Implants Res. 2019 Dec;30(12):1250-1258. doi: 10.1111/clr.13549. Epub 2019 Oct 28. PMID 31610069
- [Background] Mizumoto RM, Yilmaz B, McGlumphy EA Jr, Seidt J, Johnston WM. Accuracy of different digital scanning techniques and scan bodies for complete-arch implant-supported prostheses. J Prosthet Dent. 2020 Jan;123(1):96-104. doi: 10.1016/j.prosdent.2019.01.003. Epub 2019 Apr 27. PMID 31040026
- [Background] Dohiem MM, Abdelaziz MS, Abdalla MF, Fawzy AM. Digital assessment of the accuracy of implant impression techniques in free end saddle partially edentulous patients. A controlled clinical trial. BMC Oral Health. 2022 Nov 12;22(1):486. doi: 10.1186/s12903-022-02505-7. PMID 36371189